CLINICAL TRIAL: NCT07401771
Title: Exercise Cardiovascular Magnetic Resonance In Heart Failure With Preserved Ejection Fraction
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Barry Borlaug, Principal Investigator, Mayo Clinic
Other Study IDs: 25-012029
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Heart Failure With Preserved Ejection Fraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HFpEF (Heart Failure with Preserved Ejection Fraction)
  Interventions: Diagnostic Test: Exercise Cardiovascular Magnetic Resonance
- Non-cardiac dyspnea
  Interventions: Diagnostic Test: Exercise Cardiovascular Magnetic Resonance
- Healthy Volunteers
  Interventions: Diagnostic Test: Exercise Cardiovascular Magnetic Resonance

INTERVENTIONS:
Diagnostic Test: Exercise Cardiovascular Magnetic Resonance — Exercise Cardiovascular Magnetic Resonance is a non-invasive imaging technique that combines cardiovascular magnetic resonance (CMR) with exercise stress testing.

SUMMARY:
The purpose of this study is to internally validate low-field Ex-CMR as a noninvasive tool for diagnosing, phenotyping, and risk stratifying HFpEF in patients with exertional dyspnea.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained
2. Three groups will be enrolled:

   1. HFpEF (cardiologist-adjudicated diagnosis as verified by PI, EF≥50%)
   2. Non-cardiac dyspnea (patients have dyspnea but were found on invasive exercise testing not to have HFpEF).
   3. Healthy volunteers with no history of dyspnea or effort intolerance.

Exclusion Criteria:

1. Contraindication for low-field CMR, as indicated in MRI safety screening checklist (Research Document #1)
2. Patient inability or unwillingness to undergo Ex-CMR
3. Cardiac implants, mechanical or biological valve, causing artifacts that compromise the quality of data
4. Hospitalization for heart failure in the preceding 30 days.
5. Large R-R interval variation, caused by frequent premature ventricular contractions or non-sinus rhythms such as persistent atrial fibrillation, which, in the opinion of the investigators, compromises the quality of data acquisition, image analysis and disrupts the consistency of the cohorts
6. Myocardial infarction or unstable angina pectoris
7. Planned coronary, carotid, or peripheral artery revascularization
8. Other causes of dyspnea as indicated in patients' medical history based upon the opinion of the PI, such as restrictive cardiomyopathy or infiltrative conditions (e.g., amyloidosis), hypertrophic obstructive cardiomyopathy, primary pulmonary arterial hypertension, more than moderate chronic obstructive pulmonary disease, right heart failure due to pulmonary disease, complex congenital heart disease, severe anemia, or more than moderate mitral or aortic heart valve disease).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be identified from Mayo Clinic Cardiac Cath lab appointment lists.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Number of heart failure hospitalizations | Baseline
  Number of heart failure hospitalizations will be determined by the number of patients admitted to the hospital due to heart failure complications.
Number of cardiac deaths | Baseline
  The number of cardiac deaths will include all patients whose death is attributable to a cardiac cause.

SECONDARY OUTCOMES:
Number of deaths | Baseline
  The number of deaths will include all patient deaths, regardless of cause.

CONTACTS AND LOCATIONS:
Overall Officials: Barry Borlaug, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No